CLINICAL TRIAL: NCT05712967
Title: Role of the Host Microbiota and Il-17 in Favoring Multiple Myeloma Progression
Acronym: MICRO-MM
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Matteo Bellone, MD, MD, IRCCS San Raffaele
Other Study IDs: Observational study
Record Dates: First submitted 2022-12-23; First posted 2023-02-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolation of plasma and cells from human blood and bone marrow samples. Feces samples collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PATIENTS WITH MM: patients fulfilling the International Myeloma Working Group (IMWG) diagnostic criteria for MM
- PATIENTS WITH sMM: patients fulfilling the International Myeloma Working Group (IMWG) diagnostic criteria for SMM
- Controls: healthy controls

SUMMARY:
Goal of this observational, non-interventional study is to demonstrate that in humans a correlation exists between bone marrow (BM) levels of the cytokine interleukin 17 (IL-17) and composition of the gut microbiota in patients affected by smoldering multiple myeloma (SMM) or multiple myeloma (MM).

Enrolled SMM/MM patients will be analyzed for their bone marrow levels of IL-17 together with the distribution of T helper 17 lymphocytes in their BM and peripheral blood. These analyses will be correlated with analyses of the patients' gut microbiome to identify commensal bacteria potentially involved in Th17 cell expansion.

DETAILED DESCRIPTION:
Each year, approximately 10% of asymptomatic smoldering multiple myeloma (SMM) patients progress to incurable multiple myeloma (MM), a neoplasm of plasma cells causing anemia, bone lesions, increased blood calcium levels and renal damage. Lack of consolidated predictive biomarkers of disease progression makes the selection of SMM candidates to early treatment difficult, and a watch and wait approach is still preferred for these patients. We have recently reported results from a retrospective clinical study showing that SMM patients with higher levels of bone marrow (BM) interleukin-17 (IL-17) were at higher risk to rapidly progress to MM than SMM patients with lower IL-17 levels. Several lines of evidence in autoimmune diseases and cancer link IL-17-producing T lymphocytes (Th17) with the gut microbiota, and evidence exists in patients affected by MM that the gut microbiota impacts disease progression and susceptibility to therapies. Such link has not been investigated in patients affected by SMM.

Goal of this observational, non-interventional study is to demonstrate that in humans a correlation exists between BM levels of IL-17 and composition of the gut microbiota.

Enrolled SMM/MM patients will be analyzed for their bone marrow levels of IL-17 together with the distribution of Th17 cells in their BM and peripheral blood. These analyses will be correlated with analyses of the patients' gut microbiome to identify commensal bacteria potentially involved in Th17 cell expansion. We will seek a direct link between gut microbiota, IL-17 and MM by transplanting mice affected by MM with stool samples from the enrolled SMM/MM patients. We expect a more aggressive disease in avatar mice transplanted with stools from IL-17-high patients when compared to IL-17-low patients. Because samples will be collected both in Italy and in the USA, the study will also allow investigating the impact of additional environmental factors (e.g. Mediterranean versus high-fat diet) on host microbiota and IL-17-driven MM. Thus, primary outcome of the study will be evidence of a correlation between BM levels of IL-17 and the composition of the gut microbiota in patients affected by SMM/MM.

The recruited patients will also be monitored for disease progression or relapse after therapy. The study has no statistical power to define correlates of disease progression in these patients. However, the gut microbiome and the levels of BM IL-17 in SMM patients will be correlated to time to MM progression. Additionally, microbiome and BM IL-17 levels in MM patients eligible for hematopoietic stem cell transplantation (HSCT) will be correlated with response to the induction phase, which is routinely evaluated within 3 months. We expect better responses in patients with low levels of BM IL-17. Additionally, based on recently published experience on the role of enteric microbiome in influencing the HSCT outcomes, we have begun collecting stool samples from MM patients before and after HSCT. Therefore, once we identify patients with early relapse, we will be able to determine if they were colonized with tumor-promoting commensal bacteria following the transplant.

ELIGIBILITY:
Inclusion Criteria:

patients fulfilling the International Myeloma Working Group (IMWG) diagnostic criteria for SMM or MM, and 10 healthy controls older than 18 years and accepting to sign the informed consent

Exclusion Criteria:

* Non-Caucasian subjects.
* Subjects younger than 18 years.
* Subjects that did not accept to sign the informed consent.
* Subjects reporting infectious diseases requiring antibiotic therapy in the previous three months, ongoing antibiotic therapy or prophylaxis.
* Subjects who already underwent HSCT or under pharmacologic therapy for MM.
* Subjects affected by autoimmune diseases with the exception of thyroiditis.
* Subjects affected by HIV, HBV or HCV.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 52 patients fulfilling the International Myeloma Working Group (IMWG) diagnostic criteria for SMM or MM, and 10 healthy controls older than 18 years and accepting to sign the informed consent
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
the role of microbiota and IL17 in MM | 5YRS
  This study will provide direct evidence that the human gut microbiota modulate BM Th17 cells and MM progression . It will also provide the ground for a larger prospective clinical study on the predictive value of BM IL-17 in SMM patients.

CONTACTS AND LOCATIONS:
Overall Officials: matteo bellone, md, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anderson KC, Carrasco RD. Pathogenesis of myeloma. Annu Rev Pathol. 2011;6:249-74. doi: 10.1146/annurev-pathol-011110-130249. PMID 21261519
- [Background] Kyle RA, Larson DR, Therneau TM, Dispenzieri A, Kumar S, Cerhan JR, Rajkumar SV. Long-Term Follow-up of Monoclonal Gammopathy of Undetermined Significance. N Engl J Med. 2018 Jan 18;378(3):241-249. doi: 10.1056/NEJMoa1709974. PMID 29342381
- [Background] Rajkumar SV, Landgren O, Mateos MV. Smoldering multiple myeloma. Blood. 2015 May 14;125(20):3069-75. doi: 10.1182/blood-2014-09-568899. Epub 2015 Apr 2. PMID 25838344
- [Background] Korde N, Roschewski M, Zingone A, Kwok M, Manasanch EE, Bhutani M, Tageja N, Kazandjian D, Mailankody S, Wu P, Morrison C, Costello R, Zhang Y, Burton D, Mulquin M, Zuchlinski D, Lamping L, Carpenter A, Wall Y, Carter G, Cunningham SC, Gounden V, Sissung TM, Peer C, Maric I, Calvo KR, Braylan R, Yuan C, Stetler-Stevenson M, Arthur DC, Kong KA, Weng L, Faham M, Lindenberg L, Kurdziel K, Choyke P, Steinberg SM, Figg W, Landgren O. Treatment With Carfilzomib-Lenalidomide-Dexamethasone With Lenalidomide Extension in Patients With Smoldering or Newly Diagnosed Multiple Myeloma. JAMA Oncol. 2015 Sep;1(6):746-54. doi: 10.1001/jamaoncol.2015.2010. PMID 26181891